CLINICAL TRIAL: NCT00443599
Title: Maintaining Normal Blood Sugar Levels in Children Undergoing Heart Surgery to Reduce the Risk of Infections and Improve Recovery (The SPECS Study)
Brief Title: SPECS: Safe Pediatric Euglycemia in Cardiac Surgery
Acronym: SPECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Agus, Assistant Professor, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 512; 5R01HL088448-05 (NIH)
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Heart Defects, Congenital; Hyperglycemia
Keywords: Congenital Heart Defects; Insulin; Euglycemia; Normoglycemia
MeSH Terms: conditions — Heart Defects, Congenital; Hyperglycemia; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Experimental): Insulin was infused to target a blood glucose concentration of 80-110 mg/dL
  Interventions: Drug: Insulin
- Usual Care (Active Comparator): Insulin was infused according to the discretion of the treating clinical team.
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Insulin — Study drug is continuously infused intravenous insulin. Suggested dose is calculated by a computerized infusion algorithm using the participant's blood sugar concentration. The insulin infusion rate is titrated to maintain normal blood sugar. Participants are eligible to receive insulin while they have an in-dwelling arterial catheter.
  Other Names: Human regular insulin; Humulin R; Novolin R
  Arms: Insulin
Other: Usual Care — Participants receive standard Cardiac ICU care without tight blood glucose control.
  Arms: Usual Care

SUMMARY:
Critically ill children, including children undergoing heart surgery, commonly develop elevated blood glucose (also known as "blood sugar") levels during their illness, which can lead to poor health outcomes and an increased risk of death. This study will examine the effectiveness of maintaining normal blood glucose levels at decreasing infections and improving recovery in young children undergoing heart surgery.

DETAILED DESCRIPTION:
Children undergoing heart surgery are under significant bodily stress, which can lead to higher than normal or lower than normal blood glucose levels. A synthetic form of insulin, a naturally occurring hormone in the body, can be injected into people to normalize blood glucose levels. Insulin is most commonly used to treat people with diabetes, but it is also used in hospitals to control blood glucose levels in patients. Previous studies of adult intensive care unit (ICU) patients have shown that patients whose blood sugar levels are maintained at normal levels with the use of insulin contract fewer infections and are released more quickly from the ICU than patients who do not maintain normal blood glucose levels. This study will use a continuous blood glucose monitoring system to detect changes in blood glucose levels. Intravenous insulin infusions will be used to then safely maintain normal blood glucose levels. The purpose of this study is to determine if maintaining normal blood glucose levels during an ICU stay will help decrease the incidence of infections and improve surgical recovery in young children following heart surgery.

This study will enroll children who are undergoing heart surgery that requires a cardiopulmonary bypass procedure. Participants will be randomly assigned to either a control group or the treatment group. All participants will receive usual care while in the ICU and will undergo continuous glucose monitoring. Participants in the treatment group will receive intravenous insulin infusions to keep their blood glucose within the normal range. While in the ICU, blood will be collected from all participants once a day for the first 3 days and then once a week to monitor glucose levels, hormone levels, and measurements of nutrition and immune function. On days 1 and 5 following surgery, participants who are on a ventilator will have their breath measured to monitor heart function and energy use. Thirty days and 1 year following surgery, study researchers will contact the participant's parent or doctor to collect information on health status and any new infections at the surgical site. Children who enroll in the study will be asked to participate in follow-up neurodevelopmental evaluations at 1 and 3 years of age to assess longer term cognitive effects of tight glycemic control in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing heart surgery with cardiopulmonary bypass
* Recovering in the Cardiac ICU

Exclusion Criteria:

* Enrolled in another interventional clinical trial with related study outcomes

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 989 (Actual)
Dates: Start 2006-11; Primary Completion 2012-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Agus, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Will share with investigators based upon specific requests

REFERENCES:
- [Background] Agus MS, Javid PJ, Piper HG, Wypij D, Duggan CP, Ryan DP, Jaksic T. The effect of insulin infusion upon protein metabolism in neonates on extracorporeal life support. Ann Surg. 2006 Oct;244(4):536-44. doi: 10.1097/01.sla.0000237758.93186.c8. PMID 16998362
- [Background] Piper HG, Alexander JL, Shukla A, Pigula F, Costello JM, Laussen PC, Jaksic T, Agus MS. Real-time continuous glucose monitoring in pediatric patients during and after cardiac surgery. Pediatrics. 2006 Sep;118(3):1176-84. doi: 10.1542/peds.2006-0347. PMID 16951013
- [Background] Javid PJ, Halwick DR, Betit P, Thompson JE, Long K, Zhang Y, Jaksic T, Agus MS. The first use of live continuous glucose monitoring in patients on extracorporeal life support. Diabetes Technol Ther. 2005 Jun;7(3):431-9. doi: 10.1089/dia.2005.7.431. PMID 15929674
- [Background] Agus MS, Javid PJ, Ryan DP, Jaksic T. Intravenous insulin decreases protein breakdown in infants on extracorporeal membrane oxygenation. J Pediatr Surg. 2004 Jun;39(6):839-44; discussion 839-44. doi: 10.1016/j.jpedsurg.2004.02.013. PMID 15185208
- [Background] Gaies MG, Langer M, Alexander J, Steil GM, Ware J, Wypij D, Laussen PC, Newburger JW, Goldberg CS, Pigula FA, Shukla AC, Duggan CP, Agus MS; Safe Pediatric Euglycemia after Cardiac Surgery Study Group. Design and rationale of safe pediatric euglycemia after cardiac surgery: a randomized controlled trial of tight glycemic control after pediatric cardiac surgery. Pediatr Crit Care Med. 2013 Feb;14(2):148-56. doi: 10.1097/PCC.0b013e31825b549a. PMID 22805161
- [Result] Agus MS, Steil GM, Wypij D, Costello JM, Laussen PC, Langer M, Alexander JL, Scoppettuolo LA, Pigula FA, Charpie JR, Ohye RG, Gaies MG; SPECS Study Investigators. Tight glycemic control versus standard care after pediatric cardiac surgery. N Engl J Med. 2012 Sep 27;367(13):1208-19. doi: 10.1056/NEJMoa1206044. Epub 2012 Sep 7. PMID 22957521
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Sadhwani A, Asaro LA, Goldberg CS, Ware J, Butcher J, Gaies M, Smith C, Alexander JL, Wypij D, Agus MSD. Impact of tight glycemic control and hypoglycemia after pediatric cardiac surgery on neurodevelopmental outcomes at three years of age: Findings from a randomized clinical trial. BMC Pediatr. 2022 Sep 7;22(1):531. doi: 10.1186/s12887-022-03556-z. PMID 36071424
- [Derived] Sadhwani A, Asaro LA, Goldberg C, Ware J, Butcher J, Gaies M, Smith C, Alexander JL, Wypij D, Agus MS. Impact of Tight Glycemic Control on Neurodevelopmental Outcomes at 1 Year of Age for Children with Congenital Heart Disease: A Randomized Controlled Trial. J Pediatr. 2016 Jul;174:193-198.e2. doi: 10.1016/j.jpeds.2016.03.048. Epub 2016 Apr 23. PMID 27112038
- [Derived] Fisher JG, Sparks EA, Khan FA, Alexander JL, Asaro LA, Wypij D, Gaies M, Modi BP, Duggan C, Agus MS, Yu YM, Jaksic T. Tight Glycemic Control With Insulin Does Not Affect Skeletal Muscle Degradation During the Early Postoperative Period Following Pediatric Cardiac Surgery. Pediatr Crit Care Med. 2015 Jul;16(6):515-21. doi: 10.1097/PCC.0000000000000413. PMID 25850865
- [Derived] Agus MS, Asaro LA, Steil GM, Alexander JL, Silverman M, Wypij D, Gaies MG; SPECS Investigators. Tight glycemic control after pediatric cardiac surgery in high-risk patient populations: a secondary analysis of the safe pediatric euglycemia after cardiac surgery trial. Circulation. 2014 Jun 3;129(22):2297-304. doi: 10.1161/CIRCULATIONAHA.113.008124. Epub 2014 Mar 26. PMID 24671945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in September 2006 and ended in May 2012. All subjects received the study intervention in the Cardiac ICUs at Boston Children's Hospital (Boston, MA) and C.S. Mott Children's Hospital (Ann Arbor, MI).
Pre-assignment Details: Participants gave consent prior to cardiopulmonary bypass (CPB) surgery, randomization occurred perioperatively and initiation of the protocol occurred postoperatively. 9 subjects were removed from the study between the time of randomization and initiation of the protocol (4 for cancellation of CPB , 3 for physician decision, 2 for death).
Groups:
- Tight Glycemic Control: Insulin : Study drug is continuously infused intravenous insulin. Suggested dose is calculated by a computerized infusion algorithm using the participant's blood sugar concentration. The insulin infusion rate is titrated to maintain normal blood sugar. Participants are eligible to receive insulin while they have an in-dwelling arterial catheter.
- Standard Care: Usual Care : Participants receive standard Cardiac ICU care without tight blood glucose control.
Period: Overall Study
Arm/Group | Tight Glycemic Control | Standard Care
Started | 496 (Randomly Assigned to Tight Glycemic Control) | 493 (Randomly Assigned to Standard Care)
Completed | 490 (Included in per-protocol analysis) | 490 (Included in per-protocol analysis)
Not Completed | 6 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Death | 1 | 1
Not completed — Cardiopulmonary bypass canceled | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tight Glycemic Control | Standard Care | Total
Number analyzed (Participants) | 490 | 490 | 980
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 490 | 490 | 980
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 4.3 [1.8 to 9.7] | 4.9 [2.3 to 10.8] | 4.6 [2 to 10.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 217 | 458
  Male | 249 | 273 | 522
Region of Enrollment [Number; unit: participants]
  United States | 490 | 490 | 980

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nosocomial Infections in the Cardiac ICU
Description: Nosocomial infections that are attributable to the subject's stay in the Cardiac ICU, according to Center for Disease Control-defined criteria. These definitions are extensive and cannot be accurately condensed to fit within this space. Current CDC/NHSN criteria may be accessed through this URL: https://www.cdc.gov/nhsn/pdfs/pscmanual/17pscnosinfdef_current.pdf.
Time Frame: Measured during participant's ICU stay, a median duration of 3 days.
Measure: Number; unit: infections / 1000 pt days
Groups:
- Tight Glycemic Control: Insulin was infused to target a blood glucose concentration of 80-110 mg/dL.
  Insulin: Study drug is continuously infused intravenous insulin. Suggested dose is calculated by a computerized infusion algorithm using the participant's blood sugar concentration. The insulin infusion rate is titrated to maintain normal blood sugar. Participants are eligible to receive insulin while they have an in-dwelling arterial catheter.
- Standard Care: Insulin was infused according to the discretion of the treating clinical team.
  Usual Care: Participants receive standard Cardiac ICU care without tight blood glucose control.
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 490 | 490
infections / 1000 pt days | 8.6 | 9.9

2. Secondary Outcome: Cardiac Index (CI)
Description: Cardiac index is a measure of cardiac function, relating the cardiac output from the left ventricle in one minute to body surface area. It is calculated using the Fick principle, using oxygen consumption measured with a metabolic cart, hemoglobin levels, and the difference between arterial and superior vena cava oxygen saturation measured by co-oximetry.
Time Frame: Day 2 (day after cardiopulmonary bypass surgery).
Population: This outcome (using indirect calorimetry) was not available at the Michigan site, and not captured in Boston participants A) who had been extubated or were receiving only pressure support ventilation, B) without a properly placed catheter allowing for a true mixed venous sample or C) for whom equipment malfunction precluded an accurate measurement.
Measure: Median (Inter-Quartile Range); unit: liters/min/m^2
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 95 | 96
liters/min/m^2 | 2.0 [1.1 to 2.8] | 1.8 [1.2 to 2.6]

3. Secondary Outcome: Duration of ICU Stay
Description: Duration of ICU stay spans from post-operative cardiac ICU admission to cardiac ICU discharge.
Time Frame: The duration of cardiac ICU stay was evaluated from the date of postoperative cardiac ICU admission until the date of cardiac ICU discharge or date of death from any cause, whichever came first, assessed up to 30 days.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 490 | 490
Days | 3 [2 to 6] | 3 [2 to 6]

4. Secondary Outcome: Duration of Hospital Stay
Description: Duration of hospital stay spans from post-operative cardiac ICU admission to hospital discharge.
Time Frame: The duration of hospital stay was evaluated from the day of postoperative cardiac ICU admission until the day of hospital discharge or day of death from any cause, whichever came first, assessed up to 30 days.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 490 | 490
Days | 8 [5 to 15] | 7 [5 to 13]

5. Secondary Outcome: Duration of Endotracheal Intubation
Description: Duration of endotracheal intubation spans from endotracheal tube intubation/initiation of mechanical ventilation to endotracheal tube extubation.
Time Frame: The duration of endotracheal intubation (mechanical ventilation) was evaluated from the day of postoperative cardiac ICU admission until the day of extubation or day of death from any cause, whichever came first, assessed up to 30 days.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 490 | 490
Days | 3 [2 to 5] | 2 [1 to 5]

6. Secondary Outcome: Mortality at Hospital Discharge.
Description: Mortality is assessed at hospital discharge and at 30 days.
Time Frame: Mortality at hospital discharge (In-hospital mortality) was evaluated on the day of hospital discharge or day of death from any cause, whichever came first (no upper limit).
Measure: Number; unit: Participants
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 490 | 489
Participants | 11 | 11

7. Secondary Outcome: Mortality at 30 Days.
Description: Mortality is assessed at hospital discharge and at 30 days. If the participant is discharged from the hospital prior to 30 days, status is determined by a follow-up phone call to the family.
Time Frame: Measured at 30 days.
Population: This outcome was not measured for participants lost to follow-up at 30 days post cardiac surgery.
Measure: Number; unit: Participants
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 488 | 484
Participants | 5 | 6

8. Secondary Outcome: Cardiac Function
Description: Cardiac function is assessed by duration of vasoactive support.
Time Frame: The duration of vasoactive support was evaluated from the day of postoperative cardiac ICU admission until the last day of vasoactive support or day of death from any cause, whichever came first, assessed up to 30 days.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 490 | 490
Days | 2 [0 to 5] | 2 [0 to 5]

9. Secondary Outcome: Immune Function
Description: Immune function is assessed by C-reactive protein (CRP) on post-operative day 7.
Time Frame: Post-operative day 7.
Population: Participants analyzed include those with adequate access for blood sampling, C-reactive protein (CRP) drawn on post-operative day 7 and successful processing and preparation of samples,
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 91 | 85
mg/dL | 3.1 [1.3 to 5.6] | 4.3 [2.4 to 7.4]

10. Secondary Outcome: Endocrine Function
Description: Endocrine function is assessed by total triiodothyronine (T3) on post-operative day 7.
Time Frame: Measured during participant's ICU stay on Day 7.
Population: Thyroid hormones were assayed only if the participant remained in the cardiac ICU and there was central venous or arterial access for blood sampling.
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 90 | 81
ng/dL | 84 [60 to 122] | 75 [52 to 108]

11. Secondary Outcome: Nutritional Status
Description: Nutritional status assessed by percentage of total caloric intake as enteral nutrition during critical illness period.
Time Frame: The percentage of total caloric intake was evaluated from the day of postoperative cardiac ICU admission until the last day of the critical illness period, as defined by the presence of the arterial catheter, assessed up to 30 days.
Population: Nutritional intake was tracked during the period of critical illness, as defined by the presence of an arterial catheter.
Measure: Median (Inter-Quartile Range); unit: Percent of total caloric intake
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 397 | 393
Percent of total caloric intake | 41 [19 to 65] | 38 [11 to 66]

12. Secondary Outcome: Neurodevelopmental Evaluation, Cognitive
Description: Neurodevelopmental follow-up includes in-person testing using the Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III), measured at one year of age.
  * Bayley-III cognitive composite score ranges from 55-145, Bayley-III language composite score ranges from 47-153, and Bayley-III motor composite score ranges from 46-154.
  * Higher values indicate better neurodevelopmental outcomes.
  * These three composite scores cannot be combined and are presented as separate scores in the literature.
Time Frame: Measured at one year of age.
Population: Participants were not eligible if: born before 3/1/2008 (1 year before start of testing); age greater than one year at time of surgery; died; lived abroad; parent/guardian declined; severe disability precluded testing; did not show for testing; testing completed at greater than 18 months post eligibility.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 100 | 101
Scores on a scale | 100.2 (13.3) | 100.8 (15.6)

13. Secondary Outcome: Neurodevelopmental Evaluation, Language
Description: as for outcome 12
Time Frame: Measured at one year of age.
Population: Participants were not eligible if: born before 3/1/2008 (1 year before start of testing); age greater than one year at time of surgery; died; lived abroad; parent/guardian declined; severe disability precluded testing; did not show for testing; testing was completed at greater than 18 months post eligibility.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 100 | 101
Scores on a scale | 94.7 (13.0) | 94.7 (13.1)

14. Secondary Outcome: Neurodevelopmental Evaluation, Motor
Description: as for outcome 12
Time Frame: Measured at one year of age.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tight Glycemic Control | Standard Care
Number analyzed (Participants) | 100 | 101
Scores on a scale | 87.2 (15.8) | 88.9 (16.9)

ADVERSE EVENTS:
Time Frame: Entire course of protocol, up to 28 days
Arm/Group | Insulin | Usual Care
Serious Adverse Events (participants affected / at risk) | 16/490 | 5/490
Other Adverse Events (participants affected / at risk) | 15/490 | 19/490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin (N=490) | Usual Care (N=490)
Severe hypoglycemia (BG < 40 mg/dL) (Endocrine disorders) | 16 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin (N=490) | Usual Care (N=490)
Hypokalemia (K < 2.0 mmol/L) (Endocrine disorders) | 15 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No